CLINICAL TRIAL: NCT04349553
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel Group Dose Escalation Study to Evaluate the Safety, Tolerability and Immunogenicity of a Potential Oral Enteric Fever Vaccine (ZH9 + ZH9PA) in Healthy Participants
Brief Title: Study to Evaluate the Safety, Tolerability and Immunogenicity of a Potential Enteric Fever Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prokarium Ltd (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRK-ENT-001
Record Dates: First submitted 2020-01-11; First posted 2020-04-16 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Enteric Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Intervention Model Description: Cohort 1 will consist of 9 participants, who will receive 3 doses of 1x10^9 Colony Forming Units (CFU) of ZH9PA (6 participants) or placebo (3 participants).
  Cohort 2 will consist of 18 participants, who will receive 3 doses of 1x10^10 CFU of ZH9PA (12 participants) or placebo (6 participants).
  Cohort 3 will consist of 18 participants, who will receive 3 doses of 1x10^10 CFU of ZH9PA and 1x10^10 CFU of ZH9 (12 participants) or placebo (6 participants).
Who Masked: Participant, Investigator
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZH9PA 1x10^9 CFU (Experimental): 1mL ZH9PA 1x10^9 CFU suspension in normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  Interventions: Biological: Placebo; Biological: ZH9PA
- ZH9PA 1x10^10 CFU (Experimental): 1mL ZH9PA 1x10^10 CFU suspension in normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  Interventions: Biological: Placebo; Biological: ZH9PA
- ZH9PA 1x10^10 CFU plus ZH9 1x10^10 CFU (Experimental): 1mL ZH9PA 1x10^10 CFU suspension in normal saline and 1mL ZH9 1x10^10 CFU suspension in normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  Interventions: Biological: ZH9PA and ZH9; Biological: Placebo
- Placebo (Placebo Comparator): 1mL (Cohorts 1 and 2) or 2mL (Cohort 3) normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  Interventions: Biological: ZH9PA and ZH9; Biological: Placebo; Biological: ZH9PA

INTERVENTIONS:
Biological: ZH9PA and ZH9 — 150mL vaccine for oral administration
  Other Names: Entervax
  Arms: Placebo; ZH9PA 1x10^10 CFU plus ZH9 1x10^10 CFU
Biological: Placebo — 150mL vaccine for oral administration
Biological: ZH9PA — 150mL vaccine for oral administration
  Arms: Placebo; ZH9PA 1x10^10 CFU; ZH9PA 1x10^9 CFU

SUMMARY:
A Phase 1, randomised, double-blind, placebo-controlled, parallel group study in 45 healthy participants aged 18 to 45 years inclusive.

DETAILED DESCRIPTION:
This is a Phase I, randomised, double-blind, placebo-controlled, parallel group, single-centre study involving 45 healthy participants. The aim is to evaluate the safety and immunogenicity of Entervax, a combination vaccine against enteric fever comprising Typhi ZH9 (hereafter ZH9) plus an engineered derivative that will provide an immune response to the key antigens (LPS 0:2 and H:a flagella) from S. Paratyphi A (hereafter ZH9PA). ZH9PA has not previously been tested in humans therefore the first two cohorts comprise a dose escalation of ZH9PA and the final cohort comprises a single dose level of the combination of ZH9PA and ZH9.

ELIGIBILITY:
Inclusion Criteria:

To be confirmed at Screening

1. Healthy male and female participants 18 to 45 years of age, inclusive.
2. Female participant of childbearing potential willing to use 2 effective methods of contraception, i.e., established method of contraception + condom, if applicable (unless of non-childbearing potential or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the participant) from the first dose until 2 months after the last dose of Investigational Medicinal Product (IMP).
3. Female participant of non-childbearing potential. For the purposes of this study, this is defined as the participant being amenorrhoeic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy).
4. Female participant of childbearing potential or non-childbearing potential with a negative pregnancy test at Screening.
5. Female participant of post-menopausal status confirmed by demonstrating at Screening that the serum level of the follicle stimulating hormone (FSH) falls within the respective pathology reference range. In the event a participant's menopausal status has been clearly established (for example, the participant indicates she has been amenorrhoeic for 10 years, confirmed by medical history, etc), but serum FSH levels are not consistent with a postmenopausal status, determination of the participant's eligibility to be included in the study will be at the Investigator's discretion following consultation with the Sponsor.
6. Male participant willing to use an effective method of contraception or 2 effective methods of contraception, i.e., established method of contraception + condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the participant) from first dose until a stool sample tested for presence of the vaccine strains is negative.
7. Participant with a body mass index (BMI) of ≥ 19 or ≤34 kg/m^2 (BMI = body weight (kg) / [height (m)]^2).
8. No clinically significant history of liver or active gall bladder disease.
9. No clinically significant history of ongoing gastro-intestinal disease or abnormality.
10. No clinically significant history of previous allergy / sensitivity to ZH9/ZH9PA or sodium bicarbonate.
11. No clinically significant history of anaphylactic shock following vaccination.
12. No clinically significant history of hypersensitivity (e.g., hives/rash/swollen lips/difficulty with breathing) to azithromycin, ampicillin, trimethoprim-sulfamethoxazole or ciprofloxacin.
13. No clinically significant abnormal laboratory test results (in the opinion of the investigator) for serum biochemistry, haematology and/or urine analyses within 28 days before receiving the first dose administration of the IMP.
14. Participant with a negative urinary drugs of abuse (DOA) screen (including alcohol and cotinine) test results, determined within 28 days before the first dose administration of the IMP unless there is a documented medical explanation for the positive result other than drugs of abuse (e.g., the participant has been prescribed opioids for pain). (N.B.: A positive test result may be repeated at the Investigator's discretion).
15. Participant with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg)) and hepatitis C virus antibody (HCV Ab) test results at Screening.
16. No clinically significant abnormalities in 12-lead electrocardiogram (ECG) or vital signs determined within 28 days before first dose of IMP.
17. Participant must be available to complete the study (including all follow up visits).
18. Participant must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
19. Participant must provide written informed consent to participate in the study.

To be re-confirmed on Day 0 / prior to each dosing visit

1. Participant continues to meet all screening inclusion criteria.
2. Participant with a negative urinary drugs of abuse screen (including alcohol and cotinine) prior to dosing unless there is a documented medical explanation for the positive result other than drugs of abuse (e.g., the participant has been prescribed opioids for pain). (N.B.: A positive test result may be repeated at the Investigator's discretion).
3. Female participant of childbearing potential or non-childbearing potential with a negative pregnancy test on admission.

Exclusion Criteria:

To be confirmed at Screening:

1. Participant with any clinically significant medical (cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, autoimmune disease or current infection) or psychiatric condition (see also exclusion criterion number 21) that, in the opinion of the Investigator, precludes participation in the study. This will include any clinically significant abnormal serum biochemistry results and/or haematological results and/or urine analytical results.
2. Participant with a history of heart disease or of rheumatic fever.
3. Participant with a significant acute febrile illness (including fever of 38.0^0C or greater within 14 days) of each dose of IMP (Days 0, 21 and 42).
4. Participant who has chronic diseases: Chronic diseases will include all autoimmune and immunocompromising conditions and any other chronic condition, which at the judgment of the Investigator, may put the participant at higher risk of side effects from the study vaccine. Conditions in the latter category might include unexplained anaemia, hepato-biliary disease, uncontrolled hypertension, participant with prosthetic joints or heart valves, etc.
5. Participant with sickle cell anaemia.
6. Participant who has undertaken a course of antibiotics/antibacterials within 28 days prior to each dose of IMP (Days 0, 21 and 42).
7. Use of prescription or non-prescription drugs within 28 days or 5 half-lives (whichever is longer) prior to receiving the first dose of IMP, unless in the opinion of the Investigator and Sponsor's Responsible Physician the medication will not interfere with the study procedures or compromise participant safety.
8. Participant who uses antacids, proton pump inhibitors or H2 blockers on a regular basis or has consumed proton pump inhibitors or H2 blockers within 24 hours prior to each dose of IMP.
9. Participant who has received investigational or licensed vaccines in the 28 days prior to dosing or anticipates receiving a vaccine other than study medication up to Day 84 of the study.
10. Participant with symptoms consistent with Typhoid fever concurrent with travel to countries where typhoid infection is endemic (most of the developing world) within 2 years prior to first dose of IMP.
11. Vaccination against Typhoid within 3 years prior to first dose of IMP.
12. Ingestion of Typhoid bacteria in a challenge study within 3 years prior to dosing.
13. Participant who works as a commercial food handler.
14. Participant who is a health care worker in direct contact with patients.
15. Participant who is a childcare worker.
16. Participant who has household contact with immuno-compromised individuals, pregnant women, children < 2 years of age or individuals > 70 years of age.
17. Participant who has person(s) living with him/her who, in the opinion of the Investigator, may be at risk of disease if exposed to the vaccine strain.
18. Participant with a known impairment of immune function or receiving (or has received in the 6 months prior to study entry) cytotoxic drugs or immunosuppressive therapy (including systemic corticosteroids).
19. Participant who is a current smoker (cigarettes, tobacco and/or e-cigarettes) or has stopped smoking in the last 3 months prior to Screening.
20. A clinically significant history of drug or alcohol abuse [defined as the consumption of more than 14 units of alcohol a week] within the past two years prior to Screening.
21. Inability to communicate well with the Investigators (i.e., language problem, poor mental development or impaired cerebral function).
22. Participation in a New Chemical Entity (NCE) clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of IMP. (Washout period between studies is defined as the period of time elapsed between receiving the last dose of the previous study and receiving the first dose of the next study).
23. Donation of 450 millilitres (mL) or more blood within the 3 months before the first dose of IMP.
24. Participant who, in the opinion of the Investigator, is unsuitable for participation in the study.

To be re-confirmed at Day 0 / prior to each dosing visit:

1. Development of any exclusion criteria since the Screening visit.
2. Use of prescription or non-prescription drugs since Screening, unless in the opinion of the Investigator and Sponsor's Responsible Physician, the medication will not interfere with the study procedures or compromise participant safety.
3. Participation in a clinical study since Screening.
4. Donation of 450 mL or more blood since Screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec Research, Merthyr Tydfil, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soulier A, Prevosto C, Chol M, Deban L, Cranenburgh RM. Engineering a Novel Bivalent Oral Vaccine against Enteric Fever. Int J Mol Sci. 2021 Mar 23;22(6):3287. doi: 10.3390/ijms22063287. PMID 33807097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-six (46) subjects (45 and 1 replacement) were enrolled into the study and dosed. The study started (first visit) on 16 December 2019 and recruitment was completed by 19 June 2020.
Groups:
- ZH9PA 1x10^9 CFU: 1mL ZH9PA 1x10^9 CFU suspension in normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  ZH9PA 150mL vaccine for oral administration: Each subject received 3 doses of vaccine on Day 0, Day 21 and Day 42
- ZH9PA 1x10^10 CFU: 1mL ZH9PA 1x10^10 CFU suspension in normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  ZH9PA 150mL vaccine for oral administration: Each subject received 3 doses of vaccine on Day 0, Day 21 and Day 42
- ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU: 1mL ZH9PA 1x10^10 CFU suspension in normal saline and 1mL ZH9 1x10^10 CFU suspension in normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  ZH9PA and ZH9 150mL vaccine for oral administration: Each subject received 3 doses of vaccine on Day 0, Day 21 and Day 42
- Placebo: 1mL (Cohorts 1 and 2) or 2mL (Cohort 3) normal saline will be mixed with sodium bicarbonate 2%w/v to produce 150mL for oral administration
  Placebo 150mL vaccine for oral administration: Each subject received 3 doses of vaccine on Day 0, Day 21 and Day 42
Period: Overall Study
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Started | 7 | 12 | 12 | 15
Completed | 6 | 12 | 11 | 15
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo | Total
Number analyzed (Participants) | 7 | 12 | 12 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (3.69) | 33.0 (7.87) | 34.4 (5.81) | 36.9 (5.52) | 34.7 (6.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 7 | 3 | 18
  Male | 4 | 7 | 5 | 12 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 12 | 12 | 14 | 44
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 7 | 12 | 12 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Number of adverse events as assessed by adverse events, laboratory safety tests (biochemistry, haematology, urinalysis), vital signs and physical examination.
Time Frame: From Day 0 to Day 84
Measure: Count of Participants; unit: Participants
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 7 | 12 | 12 | 15
Participants | 4 | 9 | 8 | 9

2. Primary Outcome: Number of Participants With Abnormal Clinically or Non-clinically Significant or Out of Expected Range Tests
Description: Tests include blood pressure, heart rate, physical examination, laboratory biochemistry, haematology and urinalysis tests
Time Frame: From Day 0 to Day 84
Measure: Count of Participants; unit: Participants
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 7 | 12 | 12 | 15
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Incidence of Serious adverse events
Time Frame: From Day 85 to Day 224
Measure: Count of Participants; unit: Participants
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 7 | 12 | 12 | 15
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal Clinically or Non-clinically Significant or Out of Expected Range Tests
Description: Tests include blood pressure, heart rate, physical examination, laboratory biochemistry, haematology and urinalysis tests if these assessments are undertaken for cause.
Time Frame: From Day 85 to Day 224
Measure: Count of Participants; unit: Participants
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 7 | 12 | 12 | 15
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Fold-Increase Serum IgG Antibody Concentration of Specific Serum Immunoglobulin (Ig)G Antibodies to the Antigen H:a
Description: Fold Increase Serum IgG Antibody Concentration of specific serum immunoglobulin (Ig)G antibodies to the antigen H:a
Time Frame: Day 0, Day 21, Day 42, and Day 84
Measure: Mean (95% Confidence Interval); unit: Fold-Increase
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 6 | 12 | 11 | 15
Fold-Increase
  Day 21 | 0.984 [0.594 to 1.375] | 1.470 [1.194 to 1.746] | 1.106 [0.817 to 1.394] | 1.055 [0.808 to 1.302]
  Day 42 | 1.346 [-1.721 to 4.414] | 4.522 [2.353 to 6.691] | 1.349 [-0.917 to 3.614] | 1.119 [-0.822 to 3.059]
  Day 84 | 1.643 [-0.812 to 4.098] | 4.968 [3.232 to 6.704] | 2.417 [0.604 to 4.230] | 1.372 [-0.181 to 2.925]

6. Secondary Outcome: Fold-Increase Serum IgG Antibody Concentration of Specific Serum Immunoglobulin (Ig)G Antibodies to the Antigen H:d
Description: Fold Increase Serum IgG Antibody Concentration of specific serum immunoglobulin (Ig)G antibodies to the antigen H:d
Time Frame: Day 0, Day 21, Day 42, and Day 84
Population: The two groups did not receive the vaccine with antibodies to the antigen H:d (ZH9) so is not measured at Day 21, Day 42 or Day 84
Measure: Mean (95% Confidence Interval); unit: Fold-Increase
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 0 | 0 | 11 | 12
Fold-Increase
  Day 21 |  |  | 8.068 [6.760 to 9.376] | 0.878 [-0.374 to 2.130]
  Day 42 |  |  | 6.783 [5.731 to 7.836] | 0.838 [-0.170 to 1.846]
  Day 84 |  |  | 5.819 [4.693 to 6.946] | 0.875 [-0.204 to 1.953]

7. Secondary Outcome: Fold-Increase Serum IgG Antibody Concentration of Specific Serum Immunoglobulin (Ig)G Antibodies to the Antigen LPSO:2
Description: Fold Increase Serum IgG Antibody Concentration of specific serum immunoglobulin (Ig)G antibodies to the antigen LPSO:2
Time Frame: Day 0, Day 21, Day 42, and Day 84
Measure: Mean (95% Confidence Interval); unit: Fold-Increase
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 6 | 12 | 11 | 15
Fold-Increase
  Day 21 | 2.489 [-5.270 to 10.248] | 4.466 [-1.020 to 9.953] | 15.858 [10.127 to 21.589] | 0.964 [-3.943 to 5.872]
  Day 42 | 3.061 [-0.658 to 6.780] | 3.305 [0.675 to 5.935] | 8.877 [6.130 to 11.624] | 0.939 [-1.413 to 3.292]
  Day 84 | 2.621 [1.157 to 4.085] | 2.759 [1.723 to 3.794] | 4.386 [3.305 to 5.468] | 1.024 [0.098 to 1.950]

8. Secondary Outcome: Fold-Increase Serum IgG Antibody Concentration of Specific Serum Immunoglobulin (Ig)G Antibodies to the Antigen LPSO:9
Description: Fold Increase Serum IgG Antibody Concentration of specific serum immunoglobulin (Ig)G antibodies to the antigen LPSO:9
Time Frame: Day 0, Day 21, Day 42, and Day 84
Population: The two groups did not receive the vaccine with antibodies to the antigen LPSO:9 (ZH9) so is not measured at Day 21, Day 42 or Day 84.
Measure: Mean (95% Confidence Interval); unit: Fold-Increase
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
Number analyzed (Participants) | 0 | 0 | 11 | 12
Fold-Increase
  Day 21 |  |  | 19.292 [5.265 to 33.320] | 1.005 [-12.425 to 14.436]
  Day 42 |  |  | 11.103 [4.275 to 17.931] | 0.845 [-5.692 to 7.383]
  Day 84 |  |  | 9.686 [3.074 to 16.297] | 0.998 [-5.332 to 7.328]

ADVERSE EVENTS:
Time Frame: Up to 12 weeks post-dose (Day 84)
Arm/Group | ZH9PA 1x10^9 CFU | ZH9PA 1x10^10 CFU | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12 | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12 | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 4/7 | 9/12 | 8/12 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZH9PA 1x10^9 CFU (N=7) | ZH9PA 1x10^10 CFU (N=12) | ZH9PA 1x10^10 CFU Plus ZH9 1x10^10 CFU (N=12) | Placebo (N=15)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 3 (7) | 4 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT04349553/Prot_SAP_000.pdf